CLINICAL TRIAL: NCT02441959
Title: Full-Endoscopic vs Open Discectomy for the Treatment of Symptomatic Lumbar Herniated Disc: A Prospective Multi-Center Randomized Study
Brief Title: Full-Endoscopic vs Open Discectomy for the Treatment of Symptomatic Lumbar Herniated Disc
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator Moved Institutions
Sponsor: Yale University (Other)
Collaborators: University of New Mexico (Other); University of Washington (Other); Desert Institute for Spine Care (Unknown); Trinity Spine Center (Unknown); Baton Rouge Ortho Clinic (Unknown); Orthopedic and Neurological Consultants, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504015767
Record Dates: First submitted 2015-04-23; First posted 2015-05-12 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endoscopic Discectomy (Active Comparator): Randomized to Endoscopic Discectomy Lumbar discectomy Endoscopic Intervention type is lumbar endoscopic surgery- no device or drug
  Interventions: Procedure: Lumbar discectomy Endoscopic
- Open Discectomy (Active Comparator): Randomized to Open Discectomy Lumbar discectomy Open Intervention type is lumbar open surgery- no device or drug
  Interventions: Procedure: Lumbar discectomy Open
- Open Discectomy-Cross Over Arm (Other): Randomized to Endoscopic Discectomy Cross over to lumbar discectomy open based on surgeons assessment pre or post incision Intervention type is lumbar open surgery- no device or drug
  Interventions: Procedure: Lumbar discectomy Open

INTERVENTIONS:
Procedure: Lumbar discectomy Open — Open Discectomy
  Other Names: Intervention type is lumbar Open surgery- no device or drug
  Arms: Open Discectomy; Open Discectomy-Cross Over Arm
Procedure: Lumbar discectomy Endoscopic — Endoscopic Discectomy
  Other Names: (Intervention type is lumbar endoscopic surgery- no device or drug
  Arms: Endoscopic Discectomy

SUMMARY:
The purpose of this study is to compare the clinical and radiographic outcomes of full endoscopic lumbar discectomy versus open lumbar decompression for the treatment of lumbar herniated discs in which the patient's leg pain is greater than back pain.

DETAILED DESCRIPTION:
The study will be performed utilizing a prospective multi-center randomized model. Approximately 7 centers will be included in the study as listed above. Patients will be informed of clinical trial and asked if they would like to participate. Patients are informed that participation is optional. Patients may withdraw from study any time prior to or after surgery. Patients will be randomized 2:1 ratio endoscopic:open surgery. Both the endoscopic and open surgical techniques are utilized in standard of care. If a subject requires an open surgery approach (based on the surgeons assessment at the time of surgery pre or post incision) after they are randomized to the endoscopic arm, they will be switched to the open arm and included in the open crossover arm of the study.

Study procedures will occur at the following time points; Pre-op, 6 wk, 3 mon, 6 mon, 1 yr and 2 yr follow-up.Subjects will complete questionnaires that assess pain level and location, functional capacity, work and health status, medication usage and duration of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient equal to or greater than 18 years old.
2. Patients with single level para-central herniated discs from L1-S1.
3. VAS (Visual Analog Scale) leg > 40 mm.
4. Leg pain must be greater than back pain.
5. Minimum 6 weeks conservative treatment unless motor strength U< U4/5 and or deteriorating neurologic function.

Exclusion Criteria:

1. Lateral/subarticular, far lateral disc herniations
2. Multi-focal (multi modal) disc herniations
3. Symptomatic multiple level disc herniations
4. Active infection either spinal or otherwise
5. Prior history of lumbar spinal infection at any level
6. Spinal tumor in lumbar region
7. Dynamic (any grade) or fixed spondylolisthesis more than 3mm
8. Disc extrusion that is more superior than most inferior aspect of superior pedicle above index disc level
9. Disc extrusion that is more inferior than the middle aspect of inferior pedicle below the index disc level
10. Presence of unilateral or bilateral pars inter articularis defects (spondylolysis)
11. Disc herniation which is significantly calcified
12. Contra-lateral leg pain U>40 mm
13. History of peripheral diabetic neuropathy
14. Significant central stenosis with history of neurogenic claudication
15. Pregnancy
16. Facet cyst on symptomatic side
17. Cauda Equina syndrome past or present
18. Patients cannot have had prior lumbar surgery including IDET (Intradiscal Electrothermal Therapy) or other percutaneous surgical procedures.
19. Significant vascular claudication
20. History of radiation to the spinal column
21. History of malignancy of any type within 2 years of consideration of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Leg pain as assessed by VAS score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James J Yue, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided